CLINICAL TRIAL: NCT04186247
Title: Personalized AZithromycin/metronidAZole, in Combination With Standard Induction Therapy, to Achieve a Fecal Microbiome Community Structure and Metagenome Changes Associated With Sustained Remission in Pediatric Crohn's Disease (CD): a Pilot Study
Brief Title: Personalized AZithromycin/metronidAZole Therapy in Pediatric Crohn's Disease (CD)
Acronym: PAZAZ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The DSMB concluded that feasibility endpoints were reached in time for Week 4 but no participants receiving standard of care dietary treatment could be randomized based on the at-risk of the microbiome signature.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Crohn's and Colitis Foundation (Other); University of Amsterdam (Other); OM Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-3100; 585718 (Other Grant/Funding Number: Crohn's & Colitis Foundation)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease; Pediatric Crohns Disease
Keywords: Microbiome
MeSH Terms: conditions — Crohn Disease | interventions — Azithromycin; Metronidazole; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
  Interventions: Other: Standard of Care
- Standard of Care + Antibiotics (Experimental): SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
  Azithromycin (weeks 4-12)
  Metronidazole (weeks 4-12)
  Interventions: Drug: Azithromycin; Drug: Metronidazole; Other: Standard of Care

INTERVENTIONS:
Drug: Azithromycin — Weeks 4-12: 7.5 mg/kg azithromycin once daily (500 mg/day maximum) for five consecutive days/ week for 4 weeks, and 3 times a week for the following 4 weeks
  Other Names: Zithromax; Zmax
  Arms: Standard of Care + Antibiotics
Drug: Metronidazole — Weeks 4-12: 20 mg/kg/day of metronidazole (10 mg/kg twice daily to a maximum of 1000 mg/day) for 8 weeks
  Other Names: Flagyl
  Arms: Standard of Care + Antibiotics
Other: Standard of Care — SOC induction therapy is nutritional therapy (Crohn's disease exclusion diet + partial enteral nutrition) for up to 12 weeks. Induction therapy is as assigned by the treating gastroenterologist prior to study entry.

SUMMARY:
This is a multi-center, randomized, controlled open-label add-on design trial pilot study to evaluate the efficacy of personalized adjunctive antibiotic (azithromycin + metronidazole) therapy in pediatric subjects with mild to moderate Crohn's disease (CD) who have a microbiome profile associated with increased risk of early relapse. This an add-on design trial for subjects already receiving standard of care therapy to induce remission; there will be no placebos.

DETAILED DESCRIPTION:
The study hypothesis is that adjunctive antibiotic therapy will improve clinical response to standard of care (SOC) induction therapy in a subgroup of CD patients with a relapse-associated microbiome profile.

Prior to starting SOC induction therapy at week 0, subjects will provide a baseline stool sample that will be screened for microbiome profiles associated with risk of relapse according to an established statistical model.

At week 4, subjects with a relapse-associated microbiome will be randomized into either a control arm that will continue to receive SOC induction therapy for an additional 8 weeks, or a treatment arm that will receive adjunctive antibiotic therapy in addition to continuing to receive SOC induction therapy for an additional 8 weeks. Subjects who do not have a relapse-associated microbiome will enter a separate control arm that will continue to receive SOC induction therapy and will have data collected for exploratory objectives. Subjects who are not in clinical remission by week 4 will receive antibiotic therapy regardless of microbiome signature at baseline. Subjects will be monitored for an additional 40 weeks after the treatment period (52 weeks total).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (and assent form, as applicable);
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Male or female, aged 3 to 17 years;
4. Diagnosed with CD according to standard clinical and histological criteria, within 36 months of week 0;
5. Exhibiting mild to moderate symptoms of active disease, as determined by a Pediatric Crohn's Disease Activity Index (PCDAI) score >10 (or > 7.5 excluding the height item) and ≤37.5;
6. Fecal calprotectin level >=250 µg/g within 30 days prior to week 0 visit based on local measurement, if available, or to be arranged with lead site if an endoscopy is not performed within 30 days prior to week 0 visit.

Exclusion Criteria:

1. Current or previous use of biologic therapy;
2. Presence of stricturing, penetrating (intestinal or perianal) and/or fistulizing CD;
3. Pregnancy or lactation;
4. Have undergone intestinal resection;
5. Positive Clostridium Difficile toxin;
6. Treatment with another investigational drug or other intervention within 30 days before week 0;
7. Risk factors for arrhythmia including history of prolonged corrected QT interval (QTc), hypokalemia or hypomagnesemia, resting bradycardia, or concurrent treatment with other drugs with potential for QT prolongation;
8. History of cockayne syndrome;
9. Prior diagnosis of any hematologic condition/blood dyscrasia which may result in leukopenia (even if leukocyte count is normal at screening);
10. Known allergy or intolerance to azithromycin or metronidazole;
11. Subjects who received intravenous anti-infective within 35 days prior to week 0 visit or anti-infectives within 14 days prior to the week 0 visit;
12. Subject on oral aminosalicylates who has not been on stable doses for greater than, or discontinued within, at least 14 days prior to week 0;
13. Subject on cyclosporine, tacrolimus or mycophenolate mofetil. Stable doses (no change within 14 days prior to week 0) of azathioprine, 6-mercaptopurine or methotrexate (MTX) are not a reason for exclusion;
14. Subject who received fecal microbial transplantation within 35 days prior to week 0 visit;
15. Screening laboratory and other analyses show any of the following abnormal results:

    * aspartate transaminase (AST), alanine transaminase (ALT) > 2 X upper limit of the reference range,
    * White blood cell (WBC) count < 3.0 X 109/L,
    * Total bilirubin >= 20 micromol/liter (1.17 mg/dL); except for subjects with isolated elevation of indirect bilirubin relating to Gilbert syndrome,
    * Estimated glomerular filtration rate (GFR) by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula of < 30 mL/min/1.73 m²,
    * Hemoglobin < 80 gram/liter,
    * Platelets < 100,000/µL.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan E Van Limbergen, MD, PhD, Principal Investigator — Amsterdam UMC; Arie Levine, MD, Study Chair — Edith Wolfson Medical Centre, Tel Aviv; Francisco Sylvester, MD, Study Chair — University North Carolina
Locations (5):
- United States (2):
  - UCSF Benioff Children's Hospital, San Francisco, California
  - University of Pittsburgh Medical Center, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- IWK Health Centre, Halifax, Canada
- Wolfson Medical Centre, Tel Aviv, Israel
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina.
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with University of North Carolina.

REFERENCES:
- [Derived] Verburgt CM, Dunn KA, Otley A, Heyman MB, Verstraete S, Sunseri W, Sylvester F, de Meij T, Comeau A, Langille M, de Jonge WJ, Benninga MA, Van Limbergen JE. Personalised azithromycin+metronidazole (PAZAZ), in combination with standard induction therapy, to achieve a faecal microbiome community structure and metagenome changes associated with sustained remission in paediatric Crohn's disease (CD): protocol of a pilot study. BMJ Open. 2023 Feb 1;13(2):e064944. doi: 10.1136/bmjopen-2022-064944. PMID 36725090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen children were enrolled in the study to assess microbiome by Week 4. All participants received standard of care.
Pre-assignment Details: Of the 13 included children, 12 had microbiome data available by Week 4. One participant refused to continue SOC diet treatment and dropped out 1 week after starting.
  Three (23%) were predicted to be non-responders based on their baseline microbiome. Of these, 2 of 3 had a primary non-response to Standard of Care (SOC) treatment and did not reach clinical remission within 4 weeks.
  Ten participants were predicted to be responders. No participants were randomized.
Groups:
- Standard of Care: All participants received standard of care during the first four weeks.
- High Risk for Relapse (Group A1): SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
  Standard of Care: SOC induction therapy is nutritional therapy (Crohn's disease exclusion diet + partial enteral nutrition) for up to 12 weeks. Induction therapy is as assigned by the treating gastroenterologist prior to study entry.
- High Risk for Relapse Standard of Care + Antibiotics (Group A2); No Remission Independent of Microbiome + Antibiotics: SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
  Azithromycin (weeks 4-12)
  Metronidazole (weeks 4-12)
  Azithromycin: Weeks 4-12: 7.5 mg/kg azithromycin once daily (500 mg/day maximum) for five consecutive days/ week for 4 weeks, and 3 times a week for the following 4 weeks
  Metronidazole: Weeks 4-12: 20 mg/kg/day of metronidazole (10 mg/kg twice daily to a maximum of 1000 mg/day) for 8 weeks
  Standard of Care: SOC induction therapy is nutritional therapy (Crohn's disease exclusion diet + partial enteral nutrition) for up to 12 weeks. Induction therapy is as assigned by the treating gastroenterologist prior to study entry.
- Normal Risk for Relapse Standard of Care (Group B): SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
Period: Standard of Care (Week 0 to Week 4)
Arm/Group | Standard of Care | High Risk for Relapse (Group A1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) | Normal Risk for Relapse Standard of Care (Group B) | No Remission Independent of Microbiome + Antibiotics
Started | 13 | 0 | 0 | 0 | 0
Completed | 11 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Period: Microbiome Result at Week 4/5
Arm/Group | Standard of Care | High Risk for Relapse (Group A1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) | Normal Risk for Relapse Standard of Care (Group B) | No Remission Independent of Microbiome + Antibiotics
Started (Of the 13 included children, 12 had microbiome data available by Week 4. One participant had microbiome results available at Week 5.) | 2 | 0 | 0 | 8 | 3
Completed | 2 | 0 | 0 | 8 | 3
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Randomization/Ongoing SOC/Antibiotics
Arm/Group | Standard of Care | High Risk for Relapse (Group A1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) | Normal Risk for Relapse Standard of Care (Group B) | No Remission Independent of Microbiome + Antibiotics
Started | 0 | 0 | 0 | 8 | 3
Completed | 0 | 0 | 0 | 2 (Two children continued with standard of care until Week 52. Six others escalated to medical therapy as prescribed by their treating physician or refused to continue dietary therapy.) | 1 (One child received antibiotics and continued in the study until Week 52. One child was excluded from the study because no azithromycin suspension was available and one child received antibiotics but escalated to medical therapy by Week 10.)
Not Completed | 0 | 0 | 0 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk for Relapse (Group A1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) | Normal Risk for Relapse Standard of Care (Group B) | No Remission Independent of Microbiome + Antibiotics | Total
Number analyzed (Participants) | 1 | 2 | 9 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 9 | 1 | 13
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 6 | 1 | 7
  Male | 1 | 2 | 3 | 0 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 1 | 2 | 9 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Remission
Description: Participants stratified based on carriage of an at-risk microbiome without need for re-induction for clinical flare (new course of nutritional therapy, need to restart steroids), steroid dependence, biologic (e.g. anti-TNF) use, and/or intestinal surgery.
Time Frame: Week 52
Population: No children carrying an at-risk microbiome achieved remission by Week 4; therefore, no participants were eligible for randomization and thus these data were not collected. Only participants who remained in the study until Week 52 are reported. The other participants either refused to continue dietary therapy or needed additional medical therapy in the course of the 52 weeks due to disease activity.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care + Antibiotics: SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
  Azithromycin (weeks 4-12)
  Metronidazole (weeks 4-12)
  Azithromycin: Weeks 4-12: 7.5 mg/kg azithromycin once daily (500 mg/day maximum) for five consecutive days/ week for 4 weeks, and 3 times a week for the following 4 weeks
  Metronidazole: Weeks 4-12: 20 mg/kg/day of metronidazole (10 mg/kg twice daily to a maximum of 1000 mg/day) for 8 weeks
  Standard of Care: SOC induction therapy is nutritional therapy (Crohn's disease exclusion diet + partial enteral nutrition) for up to 12 weeks. Induction therapy is as assigned by the treating gastroenterologist prior to study entry.
Arm/Group | Standard of Care | Standard of Care + Antibiotics
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

2. Primary Outcome: Feasibility of Multinational Microbiome-randomized Trial
Description: The number of participants with microbiome data available at Week 4/5.
Time Frame: Week 4/5
Population: Two participants provided microbiome data at Baseline but did not continue after Week 1. No participants were randomized into Group A1 or Group A2. Eight participants continued SOC in Group B and three participants were eligible for antibiotics based on microbiome data and not achieving remission in Group C (two participants received antibiotics).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | High Risk for Relapse (Group A1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) | Normal Risk for Relapse Standard of Care (Group B) | No Remission Independent of Microbiome + Antibiotics
Number analyzed (Participants) | 2 | 0 | 0 | 8 | 3
Participants | 2 |  |  | 8 | 3

3. Secondary Outcome: Number of Participants With Normal Pediatric Crohn's Disease Activity Index (PCDAI) Score at Week 52
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's Disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, examination of abdomen, perirectal disease, and extraintestinal manifestations. Scores range from 0 to 100, with higher scores indicating greater disease activity.
Time Frame: Week 52
Population: No children carrying an at-risk microbiome achieved remission by Week 4; therefore, no participants were eligible for randomization and thus these data were not collected. Only 3 participants were maintained in the study until Week 52, the other participants either refused to continue dietary therapy or needed additional medical therapy in the course of the 52 weeks due to disease activity.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Antibiotics
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

4. Secondary Outcome: Number of Participants With Normal Fecal Calprotectin Levels in Stool at Week 52
Description: Fecal calprotectin is a non-invasive surrogate protein marker for bowel inflammation. The normal range is <200 mcg/g.
Time Frame: Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Antibiotics
Number analyzed (Participants) | 2 | 1
Participants | 1 | 1

5. Secondary Outcome: Number of Participants With Normal C-Reactive Protein (CRP) Levels in Blood at Week 52
Description: CRP is a blood protein marker of inflammation. CRP levels are classified as 'normal/low' or 'elevated/high' based on standard laboratory reference ranges.
Time Frame: Week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Standard of Care + Antibiotics
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

6. Secondary Outcome: IMPACT-III Score at Week 52
Description: The IMPACT III questionnaire is a 35-item assessment of health-related quality of life in patients with inflammatory bowel disease (Crohn's disease [CD] or ulcerative colitis). In this study, participants aged 9 and older will complete this questionnaire at week 0, 12, 24, and 52. Participants mark an option from 1 to 5 for each item.The total scores range from 35 to 175, with higher scores representing a better quality of life.
Time Frame: Week 52
Population: No children carrying an at-risk microbiome achieved remission by Week 4. Consequently, no participants were eligible for randomization, and these data were not collected. Additionally, no questionnaires were completed at Week 52 for any participants. Although three children continued participation through Week 52, they were not asked to complete the IMPACT-III questionnaire after the DSMB decision to stop the study.
Arm/Group | Standard of Care | Standard of Care + Antibiotics
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent until study conclusion (up to 52 weeks).
Groups:
- No Remission Independent of Microbiome + Antibiotics (Group C): SOC induction (nutritional therapy) for up to 12 weeks, as assigned by the treating gastroenterologist prior to study entry.
  Azithromycin (weeks 4-12) Metronidazole (weeks 4-12) Azithromycin: Weeks 4-12: 7.5 mg/kg azithromycin once daily (500 mg/day maximum) for five consecutive days/ week for 4 weeks, and 3 times a week for the following 4 weeks Metronidazole: Weeks 4-12: 20 mg/kg/day of metronidazole (10 mg/kg twice daily to a maximum of 1000 mg/day) for 8 weeks Standard of Care: SOC induction therapy is nutritional therapy (Crohn's disease exclusion diet + partial enteral nutrition) for up to 12 weeks. Induction therapy is as assigned by the treating gastroenterologist prior to study entry.
Arm/Group | High Risk for Relapse (Group A1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) | Normal Risk for Relapse Standard of Care (Group B) | No Remission Independent of Microbiome + Antibiotics (Group C)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/9 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 2/2 | 2/9 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk for Relapse (Group A1) (N=1) | High Risk for Relapse Standard of Care + Antibiotics (Group A2) (N=2) | Normal Risk for Relapse Standard of Care (Group B) (N=9) | No Remission Independent of Microbiome + Antibiotics (Group C) (N=1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Change in taste (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Elevated Liver Enzymes (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dilated Bile Duct (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT04186247/Prot_SAP_000.pdf